CLINICAL TRIAL: NCT02116868
Title: Usefulness of Pupillary Reflex on Remifentanil and Morphine Consumption During Laparoscopic Surgery. A Bicentric, Prospective, Randomized, Controlled Trial.
Brief Title: Pupillary Reflex Measurement to Guide Intraoperative Analgesia During Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-A01002-43
Record Dates: First submitted 2014-04-10; First posted 2014-04-17 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Scheduled Laparoscopic Surgery
Keywords: Pupillometry; Pupillary reflex; Analgesia; Laparoscopic surgery; Total intravenous anesthesia; Target controlled infusion
MeSH Terms: conditions — Agnosia | interventions — esmolol; Nicardipine; urapidil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pupillometry guided analgesia (PP) (Experimental): Analgesia is guided by pupillary reflex. The anesthesiologist in charge must adjust the peroperative remifentanil dose (Target controlled infusion) during surgery according to the algorithm proposed. Administration of antihypertensive drugs or vasopressors is also guided.
  Interventions: Device: Pupillometry guided analgesia (PP); Drug: Tailored remifentanil controlled infusion; Drug: Tailored antihypertensive drug administration
- Standard practice (ST) (No Intervention): Anesthesia and analgesia is left to the discretion of the anesthesiologist in charge. The anesthesiologist is blinded to the results of pupillometry.

INTERVENTIONS:
Device: Pupillometry guided analgesia (PP) — Analgesia is guided by pupillary reflex provided by the pupillometer (AlgiScan). The anesthesiologist in charge must adjust the peroperative remifentanil dose (Target controlled infusion) during surgery according to the algorithm proposed (Tailored remifentanil controlled infusion). Administration of antihypertensive drugs or vasopressors is also guided.
  Other Names: Algiscan Neurolight; Pupillometer
  Arms: Pupillometry guided analgesia (PP)
Drug: Tailored remifentanil controlled infusion — The anesthesiologist in charge must adjust the peroperative remifentanil dose (Target controlled infusion) during surgery according to the algorithm proposed
  Other Names: Traget controlled infusion; TCI
  Arms: Pupillometry guided analgesia (PP)
Drug: Tailored antihypertensive drug administration — Administration of antihypertensive drugs or vasopressors is guided by the results of the pupillary reflex.
  Other Names: Esmolol; Nicardipine; Urapidil
  Arms: Pupillometry guided analgesia (PP)

SUMMARY:
The purpose of this study is to determine whether analgesia guided by pupillary reflex during laparoscopic surgery is effective in opioid sparing (intraoperative remifentanil and postoperative morphine).This is a prospective, randomized, controlled study performed in two centers.

DETAILED DESCRIPTION:
For now, intraoperative analgesia remains hard to assess in the absence of reliable and validated analgesia monitor. The analysis of pupillary reflex is a new tool to assess analgesia during the intraoperative and postoperative period.

During laparoscopic surgery, carbon dioxide insufflation that produce pneumoperitoneum may induce hemodynamics events such as tachycardia or hypertension. These events may be misleading or confusing. Actually, these events are mainly considered as insufficient analgesia. Thus, anesthesiologists deepen analgesia and/or anesthesia by increasing concentration of anesthetics or opioids. These inappropriate actions may induce hypotension and/or bradycardia especially in elderly patients. On the contrary, insufficient analgesia may exist in hypovolemic patients or in patients with neuromuscular blocking agents.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists status 1 to 4
* Scheduled laparoscopic surgery
* Standardized anesthesia (TCI)
* Social security affiliation

Exclusion Criteria:

* Age < 18 yrs old
* Emergency
* BMI ≥ 35 kg.m-2
* Refusal of consent
* History of ocular pathology
* Intake of: metoclopramide, droperidol, opioids or substitutive therapies
* Patient with chronic pain
* Neurologic impairments
* Neuropathic pain
* Drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-03; Primary Completion 2018-03 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Peroperative Remifentanil consumption | From the start of anesthesia to the end of surgery (<10 hours)

SECONDARY OUTCOMES:
Number of hemodynamic events (hypertension, hypotension, tachycardia or bradycardia...) | From the start of anesthesia to the end of surgery (<10 hours)
Use of antihypertensive agents or vasopressors | From the start of anesthesia to the end of surgery (<10 hours)
Volume of fluid replacement | From the start of anesthesia to the end of surgery (<10 hours)
Pain scores | In the immediate postoperative period (<4 hours)
  Using verbal rating scale
Incidence of postoperative nausea and vomiting (PONV) | In the immediate postoperative period (<4 hours)
Time from extubation between the end of surgery and PACU admission | In the immediate postoperative period (<4 hours)
Length of stay in PACU | From PACU admission to an ALDRETE score of 10 (< 4 hours)
Immediate postoperative morphine consumption | During postanesthetic care unit (PACU) stay (<4 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Claude MEISTELMAN, MD., PhD., Study Chair — Department of Anesthesiology and Critical Care Medicine, CHU NANCY Brabois, FRANCE; Philippe GUERCI, MD, Principal Investigator — Department of Anesthesiology and Critical Care Medicine, CHU NANCY Brabois, FRANCE; Florence VIAL, MD, Principal Investigator — Department of Anesthesiology, Maternité Régionale Universitaire, CHU NANCY, France; Hervé BOUAZIZ, MD., PhD., Study Chair — Department of Anesthesiology, Maternité Regionale Universitaire, CHU NANCY, FRANCE
Locations (2):
- France (2):
  - Maternité Régionale Universitaire (MRU), Nancy, Lorraine
  - Centre Hospitalier Universitaire, Brabois, Nancy, Lorraine

REFERENCES:
- [Derived] Guerci P, Jay G, Arnout C, Herbain D, Baka N, Poirel O, Novy E, Bouaziz H, Vial F. Effects of pupillary reflex dilation-guided opioid administration on remifentanil and morphine consumption during laparoscopic surgery: A randomised controlled trial. Eur J Anaesthesiol. 2021 Sep 1;38(9):975-984. doi: 10.1097/EJA.0000000000001491. PMID 33913678